CLINICAL TRIAL: NCT06997588
Title: Study Assessing the Efficacy, Safety and Pharmacokinetics of Alpelisib in Pediatric and Adult Patients With PIK3CA-related Overgrowth Spectrum (PROS)
Brief Title: EPIK-P4: A Phase II Single-arm Study to Assess the Efficacy, Safety and Pharmacokinetics of Alpelisib (BYL719) in Pediatric and Adult Patients With PIK3CA-related Overgrowth Spectrum (PROS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719F12202; 2024-519960-42-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: PIK3CA-related Overgrowth Spectrum (PROS)
Keywords: PIK3CA-related overgrowth spectrum (PROS); Alpelisib (BYL719); Phase II; Adult; Pediatric; Adolescent
MeSH Terms: interventions — Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Adult participants ≥18 years of age.
  Interventions: Drug: Alpelisib
- Group 2 (Experimental): Children and adolescents 2 to <18 years of age.
  Interventions: Drug: Alpelisib

INTERVENTIONS:
Drug: Alpelisib — Oral Film-Coated Tablet (FCT):
  * Group 1: 250 mg once daily
  * Group 2, 6 to <18 years: 125 mg once daily (starting dose)
  Granules:
  • Group 2, 2 to <6 years: 50 mg once daily (starting dose)
  Other Names: BYL719

SUMMARY:
This study is designed to demonstrate the efficacy and assess safety and tolerability of oral daily alpelisib in participants with PIK3CA-related overgrowth spectrum (PROS).

DETAILED DESCRIPTION:
The study consists of a screening period of up to 42 days, a core period of 48 weeks and an extension period of up to 2 years to assess the efficacy, safety and pharmacokinetic (PK) of alpelisib in pediatric and adult participants with PROS.

Screening Period: Potential participants will be assessed for eligibility and undergo a whole body MRI scan to evaluate PROS-related lesions. Only those who meet all inclusion criteria will be eligible for randomization.

Core Period: Baseline is defined as the last available evaluation prior to the first dose of study treatment. Participants in Group 1 and Group 2 will be enrolled and treated with alpelisib in an open-label fashion.

* Group 1 (adults): will start with 250 mg once daily, with no dose escalation allowed.
* Group 2 (children and adolescents): will start with 50 mg once daily for participants aged 2 to <6 years, and 125 mg once daily for participants aged 6 to <18 years.

Extension 1 Period: Participants in both groups will continue their treatment under the same rules as the core period. This period will last until Week 168 following the completion of the core period for each participant. Those who complete this period before the end of the study will transition to the Extension 2 period.

Extension 2 Period: Participants will continue their treatment under the same rules as the core and Extension 1 periods until the last participant completes the Extension 2 period. Participants still deriving clinical benefit from alpelisib at the end of the study may receive post-trial access (PTA) to alpelisib.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female participants aged ≥2 years at the time of informed consent/assent.
2. Participants with diagnosis of PROS (according to Clinical Diagnostic Criteria for PROS proposed by Keppler Noreuil et al 2014) with symptomatic AND progressive overgrowth, who have syndromic disease or isolated features (with the exception of isolated macrodactyly, macrocephaly or epidermal nevus) at the time of informed consent/assent.
3. Documented evidence of a somatic mutation(s) in the PIK3CA gene performed in local laboratories using a DNA-based test AND available archival tissue (if archival tissue sample is not available, a fresh biopsy should be performed, if it is not clinically contraindicated) at the time of informed consent/assent.
4. Karnofsky (in participants >16 years of age at study entry) or Lansky (≤16 years of age at study entry) performance status index ≥50.
5. PGI-S score of mild, moderate, severe, or very severe at screening.
6. Adequate bone marrow and organ function.
7. Presence of at least 1 PROS-related measurable lesion (longest diameter ≥2 cm) confirmed by BIRC assessment and associated with complaints, clinical symptoms or functional limitations affecting the participant's everyday life.

Key Exclusion Criteria:

1. Participant with only isolated macrodactyly, epidermal nevus/nevi and macroencephaly (the only clinical feature or a combination of any of three of them), in absence of other PROS-related lesions at the time of informed consent/assent.
2. Previous treatment with alpelisib and/or any other phosphatidylinositol 3-kinase (PI3K) inhibitor(s) (except treatment attempt, defined as the attempt to treat PROS with any of PI3K inhibitors, with treatment duration less than 2 weeks and stopped at least 4 weeks prior to the first dose of study medication with alpelisib).
3. Debulking or other major surgery performed within 3 months at the time of informed consent/assent.
4. Radiation exposure for PROS treatment purpose within 12 months prior to informed consent/assent.
5. Clinically meaningful PROS-related thrombotic event (Grade 2 and more as per CTCAE v4.03) within 30 days before informed consent/assent, and/or sclerotherapy/embolization for vascular complications performed within 6 weeks before informed consent/assent.
6. Clinically meaningful bleeding from PROS-related lesion (Grade 2 and more as per CTCAE v4.03) within 30 days before study treatment initiation.
7. Participants with clinically significant worsening of PROS-related laboratory abnormalities, physical signs and symptoms (such as, but not limited to increase of D-dimers, worsening of underlying pain, newly occurring swelling or redness) indicating an uncontrolled condition during the screening phase.

Other inclusion/exclusion criteria may apply

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2028-08-02 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a confirmed objective response by BIRC | Up to Week 48
  Confirmed objective response is defined as achieving radiological response, confirmed by a subsequent assessment performed at least after 4 weeks. The achievement of radiological response requires ≥20% reduction from baseline in the sum of target lesion volumes (1 to 3 target lesions, assessed by Magnetic Resonance Imaging (MRI) by a blinded independent review committee (BIRC)), provided that none of the individual target lesions has ≥20% increase from nadir, and in absence of progression of non-target lesions and without new lesions.

SECONDARY OUTCOMES:
Change from baseline (as assessed by BIRC) in target lesion volume | Baseline, Week 12, Week 24, Week 48, Week 96, Week 144, Week 168, End of Treatment (last dose +< 14 day - Only for participants discontinuing on or prior to week 168)
  Change from baseline (as assessed by BIRC) in target lesion volume will be summarized descriptively
Change from baseline (as assessed by BIRC) in MRI-measurable non-target lesion volume | Baseline, Week 12, Week 24, Week 48, Week 96, Week 144, Week 168, End of Treatment (last dose +< 14 day - Only for participants discontinuing on or prior to week 168)
  Change from baseline (as assessed by BIRC) in MRI-measurable non-target lesion volume will be summarized descriptively
Change from baseline (as assessed by BIRC) in all MRI-measurable (target and non-target) lesion volume | Baseline, Week 12, Week 24, Week 48, Week 96, Week 144, Week 168, End of Treatment (last dose +< 14 day - Only for participants discontinuing on or prior to week 168)
  Change from baseline (as assessed by BIRC) in all MRI-measurable (target and non-target) lesion volume will be summarized descriptively
Change from baseline (as assessed by BIRC) in other non-target lesion | Baseline, Week 12, Week 24, Week 48, Week 96, Week 144, Week 168, End of Treatment (last dose +< 14 day - Only for participants discontinuing on or prior to week 168)
  Change from baseline (as assessed by BIRC) in other non-target lesion will be summarized descriptively
Appearance of new lesions (as assessed by BIRC) | Week 12, Week 24, Week 48, Week 96, Week 144, Week 168, End of Treatment (last dose +< 14 day - Only for participants discontinuing on or prior to week 168)
  Appearance of new lesions (as assessed by BIRC) will be summarized descriptively
Proportion of participants with a radiological response | Week 12, Week 24, Week 48, Week 96, Week 144, Week 168, End of Treatment (last dose +< 14 day - Only for participants discontinuing on or prior to week 168)
Duration of Response (DoR) | From first documented response until progression of PROS lesions or death, assessed up to approximately 3 years
  Duration of response (DOR) is defined as the time from the first documented confirmed objective response until progression of any PROS lesion by BIRC or death or rescue surgery for any PROS lesion.
Alpelisib plasma concentration | Week 1 Day 1 (Post-dose 3 hour), Week 4 Day 1 (Pre-dose and Post-dose 3 hour), Week 12 Day 1 (Pre-dose and Post-dose 3 hour)
Change from Baseline in Brief Pain Inventory (BPI) | Baseline, Week 4, Week 8, Week 12, Week 16, Week 24, Week 48, Week 72, Week 96, Week 120, Week 144, Week 168, End of Treatment (last dose +< 14 days)
  Two items from the Brief Pain Inventory (BPI) will be used for adult and pediatric participants aged 12 years and older. The first item assesses the worst pain intensity in the past 24 hours, with responses on an 11-point scale from 0 (no pain) to 10 (pain as bad as you can imagine). The second item evaluates pain interference with general activity in the past 24 hours, also on an 11-point scale from 0 (does not interfere) to 10 (completely interferes).
Change from Baseline in Wong-Baker Faces Scale | Baseline, Week 4, Week 8, Week 12, Week 16, Week 24, Week 48, Week 72, Week 96, Week 120, Week 144, Week 168, End of Treatment (last dose +< 14 days)
  For children aged 3-11 years, the Wong-Baker FACES® Pain Rating Scale will be used instead of the BPI worst pain intensity question. This scale features six faces showing increasing levels of pain, each with a numeric rating and a descriptor (from 0 'no hurt' to 10 'hurts worst'). Children will select the face that best represents their pain level. There is no pain intensity scale for children under 3 years.
Change from Baseline in Patient Global Impression of Symptom Severity (PGI-S) | Baseline, Week 4, Week 8, Week 12, Week 16, Week 24, Week 48, Week 72, Week 96, Week 120, Week 144, Week 168, End of Treatment (last dose +< 14 days)
  A Patient Global Impression of Symptom Severity (PGI-S) item will be used to understand the overall severity of symptoms experienced and clinical meaningfulness of treatment effects experienced during this study. This item includes 5 response options: no symptoms, mild, moderate, severe, and very severe. This scale can be completed by the parent/caregiver for pediatric participants aged <12 years.
Time to Treatment Failure (TTF) | From Baseline up to approximately 3 years
  Time to Treatment Failure (TTF) is defined as the time from alpelisib treatment start date until disease progression supported by radiological assessment performed by BIRC, death, rescue surgery for any PROS lesion or discontinuation of alpelisib due to any reason other than technical problems or study termination by the sponsor. Participants who complete the study, are ongoing treatment or discontinue alpelisib due to technical problems (e.g. drug supply issues, site prematurely ends study participation) or study termination by the sponsor will be censored at the date of last study treatment received.
Overall Clinical Response | From Baseline up to approximately 3 years
  The proportion of participants with overall clinical response reported as improvement, stable or worsening of clinical condition, as assessed by the Investigator will be summarized descriptively.
Change from Baseline in symptoms and complications/comorbidities associated with PROS | From Baseline up to approximately 3 years
  Changes in symptoms and complications/comorbidities (i.e., walking impairment, cardiac/pulmonary/renal function, pain, Karnofsky/Lansky performance status) will be summarized descriptively. For each complication/comorbidity, only participants who have this reported as being present at baseline will be included in the analysis. When new symptoms/complications/comorbidities appear at any time of study therapy, they will be assessed for clinical significance and reported as adverse events when applicable.
Percentage of participants with healthcare visits/hospitalized due to PROS | Up to at least 3 years
  Percentage of participants with healthcare visit/hospitalized due to PROS will be assessed for Group 1 and Group 2.
Percentage of participants with surgeries required to manage PROS | Up to at least 3 years
  Percentage of participants requiring rescue surgery due to PROS will be assessed for Group 1 and Group 2.
Number of Adverse Events and Serious Adverse Events as assessed by CTCAE criteria | Up to at least 3 years
  Treatment emergent Adverse Event (TEAEs) in this study were events that started after the first dose of study treatment and until 30 days after the last dose of study treatment, or events present prior to the first dose of treatment which increased in severity based on preferred term within 30 days after the last study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- Washington University, St Louis, Missouri, United States
- Australia (2):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, North Adelaide, South Australia
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Ghent, Belgium
- France (4):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Tours
- Germany (5):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Berlin
- Italy (2):
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Spain (2):
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com